CLINICAL TRIAL: NCT06367075
Title: The Efficacy and Safety of Cadonilimab(AK104) With Adriamycin for First-line Treatment of Advanced Soft Tissue Sarcoma: a Multicenter, Single-arm, Phase II Clinical Trial
Brief Title: A Trial of Cadonilimab With Adriamycin in Patients With Advanced Soft Tissue Sarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Sun Yat-sen University (Other); Yunnan Cancer Hospital (Other); The Affiliated Hospital Of Guizhou Medical University (Other); First Affiliated Hospital of Guangxi Medical University (Other); Second Xiangya Hospital of Central South University (Other); Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-sarcoma-202401
Record Dates: First submitted 2024-04-10; First posted 2024-04-16 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Advanced Soft-tissue Sarcoma
Keywords: Advanced Soft-tissue Sarcoma; cadonilimab; chemotherapy; Anti-PD-1/CTLA4 bispecific antibody
MeSH Terms: interventions — Doxorubicin

STUDY DESIGN:
Intervention Model Description: cadonilimab (AK104) with adriamycin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cadonilimab (AK104) with adriamycin (Experimental): Run-In Period（C1）: cadonilimab10mg/kg, d1 ,q3w; Treatment period（C2~C7）: adriamycin 25mg/m2, d1-d3，q3w; cadonilimab 10mg/kg, d1, q3w; Maintenance period（C8~）: cadonilimab 10mg/kg, d1, q3w
  Interventions: Drug: Cadonilimab; Drug: Adriamycin

INTERVENTIONS:
Drug: Cadonilimab — injectable solution
  Other Names: AK104
Drug: Adriamycin — injectable solution
  Other Names: Doxorubicin

SUMMARY:
This is a single-arm, multicenter trial of cadonilimab (AK104) with adriamycin in patients with first-line advanced soft tissue sarcoma. the primary objective is to evaluate objective response rate of cadonilimab with adriamycin.

DETAILED DESCRIPTION:
In this study, the screening period does not exceed 28 days, and subjects who are qualified after completion of the screening examination and evaluation entered the treatment period and undergo study treatment and visits as specified in the protocol. In particular, tumor imaging assessments are performed every 2 cycles during the first 16 cycles; thereafter, tumor imaging assessments are performed every 4 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were pathologically confirmed soft tissue sarcoma (soft tissue sarcomas other than alveolar/embryonal rhabdomyosarcoma, clear cell sarcoma, extraosseous Ewing sarcoma, alveolar soft tissue sarcoma, well differentiated liposarcoma, extraosseous myxoid chondrosarcoma, etc.)
* The patient was diagnosed as progressive and the investigators determined that the lesion was not suitable for surgical treatment
* The patients had not received systemic therapy (including chemotherapy, targeted therapy and bioimmunotherapy) for advanced soft tissue sarcoma. More than 6 months have passed since the end of neoadjuvant/adjuvant therapy (including chemotherapy, targeted therapy, bioimmunotherapy, etc.), and the cumulative dose of adriamycin used in the past was ≤100 mg/m2
* In patients with measurable disease, lesions are defined and monitored by RECIST v1.1
* Aged ≥ 18 years old, < 60 years old
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1, amputees can be 0-2
* Expected survival > 3 months
* Adequate organ and bone marrow function, defined as follows: ① Blood routine (14 days before screening without blood transfusion, without G-CSF, without drug correction): neutrophil count (ANC) ≥ 1.5 × 10^9/L; platelet count (PLT) ≥ 100 × 10^9/L; hemoglobin (Hb) ≥ 100 g/L; ② Blood biochemistry: serum creatinine (Cr) ≤ 1.5 × upper limit of normal (ULN) or creatinine clearance ≥ 60ml/min; total bilirubin (TBIL) ≤ 1.5 × ULN; aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≤ 2.5 × ULN, The subjects with liver metastasis should be ≤ 5 × ULN; ③ Coagulation function: international normalized ratio (INR) ≤ 1.5, prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN; ④ Urinalysis: urine protein < 2 +; if urine protein ≥ 2 +, the 24-hour urine protein quantification must be ≤ 1g; ⑤ thyroid stimulating hormone (TSH) ≤ ULN and ≥ LLN; if abnormal, T3 and T4 levels should be investigated, normal T3 and T4 levels can be included
* Cardiac function:1) 12-lead electrocardiogram showed no severe arrhythmias, QTcF ≤ 480 ms; 2) No signs of myocardial ischemia; 3) LVEF ≥55% by cardiac ultrasound (measured by the biplane Simpson method); 4) NT-proBNP < age cutoff value; 5) Troponin within normal values.
* Agree and have signed informed consent, willing and able to comply with scheduled visits, study treatment, laboratory tests and other test procedures
* Women of childbearing potential should have a negative serum or urine pregnancy test within 72 hours prior to receiving the first dose of study treatment; and should be willing to use one acceptable contraception (i.e., oral contraceptives, condoms, intrauterine devices [IUDs]) throughout the period of taking study treatment and for at least 3 months after the last dose of study drug(s). For men, surgical sterilization or consent to appropriate contraception during observation and up to 90 days after the last treatment should be used

Exclusion Criteria:

* known allergy to recombinant humanized anti-PD-1 monoclonal antibody drugs and their components
* Known allergy to recombinant humanized anti-CTLA-4 monoclonal antibody drug and its components
* known allergy to any component of the cadonilimab formulation
* Patients with cardiac disease class II or higher as determined by the New York Heart Association (NYHA) score
* Palliative radiotherapy within 2 weeks prior to the first dose
* Other active malignancy within 5 years prior to enrollment. Except for locally curable malignancies (manifested as cured) such as basal or cutaneous squamous cell carcinoma, superficial bladder cancer, endometrial carcinoma in situ, cervical carcinoma in situ, or breast carcinoma in situ
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study
* Active autoimmune disease requiring systemic therapy within 2 years prior to the start of study treatment, or autoimmune disease that, in the judgment of the Investigator, is likely to recur or for which treatment is planned; except for the following: skin diseases not requiring systemic therapy (e.g., vitiligo, alopecia areata, psoriasis, or eczema); hypothyroidism due to autoimmune thyroiditis requiring only a stable dose of hormone replacement therapy; well-controlled type I diabetes mellitus; childhood well-controlled type I diabetes mellitus; subjects whose childhood asthma has completely resolved and does not require any intervention in adulthood; and subjects who, in the judgment of the investigator, have a disease that will not recur in the absence of external triggers
* Inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis, or chronic diarrhea) that is active or requires clinical management
* Subjects will require systemic therapy with corticosteroids (>10 mg/day of prednisone equivalents) or other immunosuppressive medications within 14 days of administration of study drug. Inhaled or topical topical steroids and adrenal replacement doses >10 mg/day of prednisone equivalent are allowed in the absence of active autoimmune disease. Topical, ocular, intra-articular, intranasal and inhaled corticosteroids (with minimal systemic absorption) are permitted in subjects. Physiologic replacement doses of systemic corticosteroids are permitted, even if >10 mg/day of prednisone equivalent. Short-term use of corticosteroids is permitted for prophylaxis (e.g., contrast allergy) or for treatment of non-autoimmune diseases (e.g., delayed hypersensitivity reactions due to contact allergens)
* Known history of positive test for human immunodeficiency virus or known acquired immunodeficiency syndrome
* History of known allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation
* Known presence or history of interstitial lung disease
* Received a live vaccine within 30 days prior to the first dose of cadonilimab or plan to receive a live vaccine during the study period
* Subjects with necrotic lesions detected on examination within 4 weeks prior to enrollment that, in the judgment of the investigator, pose a risk of major bleeding
* Serious infection, including but not limited to concomitant complications requiring hospitalization, sepsis, or severe pneumonia, within 4 weeks prior to first dose
* Known active tuberculosis (TB). Subjects suspected of having active TB will be examined by chest X-ray, sputum, and exclusion by clinical signs and symptoms
* Patients with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers with HBV DNA >1000 IU/mL, and patients with active hepatitis C should be excluded. Inactive hepatitis B surface antigen (HbsAg) carriers, treated and stabilized hepatitis B patients (HBV DNA <1000 IU/mL), and cured hepatitis C patients may be enrolled. For HCV Ab-positive subjects, participation in the study is eligible only if the HCV RNA test result is negative
* Major surgical procedure within 30 days prior to the first dose of cadonilimab or have not fully recovered from a prior procedure. Localized surgical procedures (e.g., systemic port placement, core needle biopsy, and prostate biopsy) are permitted provided that the procedure is completed at least 24 hours prior to the time of the first dose of study treatment medication
* Presence of known meningeal metastases, spinal cord compression, molluscum contagiosum disease, or active brain metastases. However, enrollment is allowed for subjects who meet the following requirements and have a measurable lesion outside the CNS: 1) previously untreated and currently asymptomatic (e.g., no neurologic deficits, seizures, or other signs and symptoms typical of CNS metastases; glucocorticoid therapy is not required); 2) asymptomatic after treatment has been imaging stable for at least 4 weeks prior to the initiation of study treatment (e.g., no new or enlarging brain metastatic lesion ) and have discontinued systemic glucocorticoid and anticonvulsant medication for at least 2 weeks
* Subjects with pleural effusions, pericardial effusions, or ascites that, in the judgment of the Investigator, remain unstably controlled using repeated drainage or other methods
* Uncontrolled co-morbidities, including symptomatic congestive heart failure (grade 3 or 4 as determined by the New York Heart Association functional classification), uncontrolled hypertension, unstable angina, poorly controlled cardiac arrhythmias, acute or evidence of ongoing myocardial ischemia, severe active peptic ulcer disease or gastritis, or mental illness/social disease that would limit the subject's ability to comply with the study requirements or interfere with the subject's ability to provide written mental illness/social condition that would limit the subject's ability to provide informed consent. Any arterial thromboembolic event, including myocardial infarction, cerebrovascular accident, or transient ischemic attack, history of deep vein thrombosis, pulmonary embolism, or any other serious thromboembolism within 6 months prior to enrollment
* Unreversed toxicity from prior antineoplastic therapy, defined as toxicity that has not returned to NCI CTCAE version 5.0 grade 0 or 1, or to a level specified in the inclusion/exclusion criteria (except alopecia areata). Subjects who experience irreversible toxicity that is not expected to worsen with administration of study drug (e.g., hearing loss) may be included in the study after consultation with the Medical Ombudsman. Subjects with radiotherapy-induced long-term toxicity that, in the judgment of the Investigator, is not reversible may be included in the study after consultation with the Medical Ombudsman
* Females who are pregnant or breastfeeding
* Any condition that, in the opinion of the Investigator, may render treatment with the study drug risky or will interfere with the evaluation of the study drug or the safety of the subject or the resolution of the study results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | from the first drug administration up to two years
  ORR is the proportion of patients with best response of complete response (CR) and partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and iRECIST

SECONDARY OUTCOMES:
Disease control rate (DCR) | from the first drug administration up to two years
  Proportion of patients whose best overall response is either CR, PR, or SD
Duration of response (DOR) | from the first drug administration up to two years
  Time from first documented response (CR or PR) until documented disease progression or death, whichever occurs first
Progression-free survival (PFS) | from the first drug administration up to two years
  Time from the date of first study treatment administration to the date of first documented tumor progression or death due to any cause, whichever occurs first
Overall survival (OS) | from the first drug administration up to two years
  Time from the date of first study treatment administration to the date of death due to any cause
Adverse event (AE) | From the subject signs the ICF to 90 days after the last dose of study treatment or initiation of other anti-tumor therapy, whichever occurs first
  To assess the safety and tolerability of cadonilimab plus adriamycin in participants with advanced soft tissue sarcoma

CONTACTS AND LOCATIONS:
Overall Officials: jing chen, doctor, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No